CLINICAL TRIAL: NCT01913626
Title: Assessing the Efficiency of Cognitive Group Therapy for Patient With Subjective Memory Complains Using the WebNeuro System From Brain Resource(BRC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC130044-13CTIL
Record Dates: First submitted 2013-07-22; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Subjective Memory Complains
Keywords: subjective memory complains

ARMS (1):
- cognitive group therapy (Experimental): patient with subjective memory complains will participate in cognitive group therapy including eight meetings of practicing cognitive strategy to improve the memory .
  Interventions: Behavioral: cognitive group therapy

INTERVENTIONS:
Behavioral: cognitive group therapy — the cognitive group therapy is composed of eight meetings including information about memory processes, learning and practicing tools and strategies to improve cognition and memory.

SUMMARY:
assessing the Efficiency of cognitive group therapy for patients with subjective memory complains, using the neuropsychological computerized assessment of WebNeuro by Brain resource (BRC).

DETAILED DESCRIPTION:
the study includes patients with subjective memory complains - who are concerned about having memory problems, that passed successfully the conventional basic cognitive assessment and who are not demented.

the patients were referred to our occupational therapy clinic for cognitive group therapy.

the aim of the study is to assess the efficiency of such therapy, using the neuropsychological computerized assessment of WebNeuro by Brain resource (BRC). the computerized assessment last 40 minutes and provide information about different cognitive aspects compared to a norm according to age, sex and education.

each patient will pass the neuropsychological computerized assessment twice: at the beginning of the study and after participating in the cognitive group therapy.

the cognitive group therapy is composed of eight meetings including information about memory processes, learning and practicing tools and strategies to improve cognition and memory.

each individual will be his one control, we will compare the patient achievements in the different cognitive aspects before and after the cognitive intervention.

our hypothesis is that the cognitive group therapy will improve the participants achievements in the neuropsychological computerized assessment.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years old and more
* 8 years of education
* know reading and writing in hebrew
* know how to use the computer

Exclusion Criteria:

* neurologic or psychiatric conditions: apraxia, aphasia, depression, brain tumor

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
the patient achievements in the different cognitive aspects assessed by the computerized neuropsychological assessment of WebNeuro by Brain resource (BRC) | 10 weeks
  the WebNeuro wellness report brings together information on diagnostic symptoms and negative feelings as well as cognitive information on self regulation, thinking and emotion (impulsivity and cognition difficulties in additional areas of thinking - attention, concentration and memory) .

CONTACTS AND LOCATIONS:
Locations (1):
- geriatric rehabilatation department , Meir medical center, Kfar Saba, Israel